CLINICAL TRIAL: NCT04930510
Title: IncIncidence and Prognosis of Coronary Artery Disease in Elderly People Over 80 Years Referred for TAVI
Brief Title: Coronary Artery Disease in Elderly People Referred for TAVI
Acronym: CEPTAVI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0208
Record Dates: First submitted 2021-05-25; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Aortic Stenosis; Coronary Ang
Keywords: Patients over 80 years; TAVI; coronary artery disease; quality of life
MeSH Terms: conditions — Aortic Valve Stenosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 : Elderly 80 years or over patients referred for TAVI with CAD: Elderly 80 years or over patients referred for TAVI with CAD Group 1: Coronary lesion defined as significant (>50% narrowing) on the coronary angiography performed before TAVI, with or without PCI (decision of the heart team) Description of the coronary lesions included: proximal/non proximal, number of lesions, location of lesion
- Group 2 : No significant coronary disease group: No significant coronary disease group in the cohort of elderly 80 years or over referred for TAVI

SUMMARY:
The investigators prognostic impact of coronary artery disease (CAD) and of percutaneous coronary intervention (PCI) in patients with indication of TAVI is controversial, particularly in elderly population where CAD and aortic stenosis (AS) are frequent and commonly coexisted. (1-2) The primary end point of this prospective study is to compare major cardiovascular event at one year of follow up in patients over 80 years with severe aortic stenosis who referred for TAVI with or without associated CAD.

The investigators will also assess (secondary endpoint) the impact of PCI on symptoms, major events and quality of life using geriatric parameters. The study will be conducted in the University hospital of Montpellier between November 2020 and November 2022

DETAILED DESCRIPTION:
Patients will be prospectively included in the study when aged of 80 years old or over and referred for TAVI at the university hospital of Montpellier.

Two groups of patients will be considered after coronary angiography which is systematic before TAVI Group 1: patients with significant > 50 % narrowing coronary stenosis ( revascularization by PCI / no revascularization) Group 2: No coronary lesion

Considering an end point at 1 year and a precision wished to i ± 6 percent with an alpha risk of 5 %, it's proposed , by the formula p= [(1.96)2 x [p(1-p)] / i2 ], a number of 170 subjects needed to highlight a incidence of major cardio-vascular event of 20 percent in the studied population.

Data collection by informatic files will include :

* Cardio vascular risk factor and medical history with evaluation of Charlston score
* Previous drug therapy
* Lifestyle : living alone or not, nursing home, ; home help
* Symptoms (angina (CSS classification) ; dyspnea (NHYA classification))
* Renal function (DFG) at admission
* Results of coronary angiography (number of lesions, proximal or non proximal, location of coronary stenosis)
* Geriatric assessment : autonomy, disability in daily living, weigh, BMI, falls, cognitive functions tests, assessment of the mood state by GDS
* Results of TAVI (success and complications of the procedure according to VARC2 criteria)
* Results of coronary revascularization if performed
* Length of hospitalisation for TAVI (days), length of stay in ICU (Intensive Care Unit) if necessary
* Events during the hospitalisation for TAVI (VARC and BARC criterias)

Follow up at 6 month (middle analysis) and at one year (primary end point) by phone conversation with the patient for assessment of :

* Major cardio-vascular events
* Hospitalisation occurred
* Short geriatric evaluation including :

  * cognition by Ottawa3DY
  * autonomy by ADL
  * polypharmacy
  * number of fall in the past 6 month
  * last weight
  * quality of life (Fried criterias)
  * mood state by GDS If neurocognitive disorders are known or discovers, data patient's validity will be check by calling his caregiver and/or his general practitioner (if caregiver not available).

Analysis associated of the computerized patient record.

ELIGIBILITY:
Inclusion criteria:

* patient aged 80 and over
* hospital admission for evaluation before TAVI indicated for symptomatic and severe aortic stenosis
* patient's consent

Exclusion criteria:

* absence of coronarography
* severe angina (class 3 or 4)
* stenosis of left main coronary artery > 50%
* stenosis of the left anterior descending artery > 90%
* decision of surgical valve replacement

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged of 80 years or over who are admitted in cardiology for TAVI
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the incidence of major cardio-vascular event | 1 year
  Comparison of the incidence of major cardio-vascular event at one year follow up in elderly 80 or over referred for TAVI with (group 1) or without CAD (group 2).
  Major cardio vascular events evaluated at 1 year follow-up include:
  * Death (total and cardiovascular)
  * ischemic stroke,
  * haemorrhagic stroke,
  * acute coronary syndrome,
  * severe angina (> class 2),
  * major bleeding or vascular complications (>BARC2),
  * Re-hospitalisation for cardiac events

SECONDARY OUTCOMES:
Incidence of CAD | 1 year
  Incidence of CAD in the elderly over 80 years old during the pre TAVI evaluation Evaluate the coronary disease impact in the elderly over 80 referred for TAVI by the number of patients over 80 years with significant coronary lesions compared to global TAVI population over 80 years
Length of hospitalisation | 1 year
  Length of hospitalisation with or without coronary disease, with or without PCI.
  Length of hospitalisation in total and in the ICU if it's happened to evaluated the economic impact of CAD and therapeutic strategy.
Rate of ischaemic | 1 year
  ischaemic event (acute coronary syndrome, severe angina)
Rate of vascular/bleeding events according to strategy of care (PCI/no PCI) | 1 year
  minor bleeding (BARC 1 and 2) and major (BARC 3 et 4) event or vascular complication (VARC 2).
Re-hospitalization for cardiac events | 1 year
  Re-hospitalization for cardiac events
Quality of life with assessment of clinical status | 1 year
  Quality of life with assessment of clinical status by geriatrics tests geriatrics tests by phone interview of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Florence Leclercq, PU PH, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Background] Cao D, Chiarito M, Pagnotta P, Reimers B, Stefanini GG. Coronary Revascularisation in Transcatheter Aortic Valve Implantation Candidates: Why, Who, When? Interv Cardiol. 2018 May;13(2):69-76. doi: 10.15420/icr.2018:2:2. PMID 29928311
- [Background] Matta AG, Lhermusier T, Parada FC, Bouisset F, Canitrot R, Nader V, Blanco S, Elbaz M, Roncalli J, Carrie D. Impact of Coronary Artery Disease and Percutaneous Coronary Intervention on Transcatheter Aortic Valve Implantation. J Interv Cardiol. 2021 Mar 24;2021:6672400. doi: 10.1155/2021/6672400. eCollection 2021. PMID 33824628